CLINICAL TRIAL: NCT07067892
Title: Effectiveness of Ultrasonography-Guided Serratus Posterior Superior Intercostal Plane Block in Thoracic Postherpetic Neuralgia: A Retrospective Cohort Study
Acronym: pain
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: postherpetic neuralgia, block
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Postherpetic Neuralgia ( PHN ), Ultrasound Guided, Block; Ultrasound Guided Injection
MeSH Terms: conditions — Neuralgia, Postherpetic; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Effectiveness of Ultrasonography-Guided Serratus Posterior Superior Intercostal Plane Block in Thora

SUMMARY:
Postherpetic neuralgia (PHN) is a chronic pain syndrome that can be resistant to treatment, leading to physical and social disability, psychological disturbances, and potentially persisting for years . The varicella-zoster virus remains latent in the sensory neurons of individuals who have previously contracted varicella (chickenpox). Reactivation of the latent virus results in herpes zoster (HZ). In most patients, HZ initially presents with dermatomal pain, and within a few days, characteristic dermatomal vesicular eruptions typically develop. These skin lesions usually heal within 2-4 weeks; however, pain may persist even after the resolution of the rash .

The pathogenesis of PHN involves increased sensitization of central neurons, decreased function of inhibitory neuronal pathways, inflammation and nerve injury within the peripheral nervous system, and abnormal signal transmission following such damage. PHN represents the most common complication of HZ. It occurs in approximately 9-19% of all patients with HZ. The incidence of PHN increases with advancing age: it affects approximately 2% of individuals younger than 50 years, about 20% of those older than 50 years, and nearly 35% of those older than 80 years . Various treatment modalities, including pharmacologic agents and interventional procedures, are available for the management of PHN-related pain. This study primarily aims to evaluate the change in pain in PHN patients who underwent SPSIPB using the NRS-11. The secondary aim was to evaluate the effect of SPSIPB on neuropathic pain characteristics using the DN-4 scale and to investigate its effects on patients' quality of life using SF-12 scale.

DETAILED DESCRIPTION:
After obtaining approval from the relevant ethics committee (University of Health Sciences, Istanbul Kanuni Sultan Suleyman Training and Research Hospital, KAEK/2025.05.139), patients over 18 years of age who underwent a single-session ultrasound (US)-guided serratus posterior superior intercostal plane block (SPSIPB) in the thoracic region (T1-T10 dermatomes) due to PHN between June 2023 and February 2025 were retrospectively evaluated. SPSIPB was performed in patients whose complaints persisted despite existing medical treatments. The study was conducted in accordance with the Declaration of Helsinki. Written informed consent was obtained from all patients enrolled in the study, which was carried out at the pain clinic of a tertiary care hospital. This retrospective, single-center cohort study was designed.

A total of 34 patients who met the inclusion criteria were included in the study .

Patients were excluded if they had cervical disc herniation; a history of trauma or surgery involving the neck, shoulder, or back; malignancy; kyphoscoliosis; a history of inflammatory diseases (e.g., rheumatoid arthritis, ankylosing spondylitis); congenital spinal anomalies; neck pain accompanied by neurological deficits; pregnancy; mental or psychotic disorders; hematologic diseases causing bleeding or coagulation disorders; use of antiplatelet or anticoagulant drugs or medications predisposing to bleeding; severe systemic infections such as sepsis; local infections at the planned intervention site; known allergies to any of the drugs to be used; or a history of invasive procedures for PHN in the thoracic region within the past 3 months.

Data Collection and Assessment Scales The following data were collected: Age, gender, body mass index (BMI), affected side in PHN, duration of PHN and affected dermatome, history of HZ vaccination (live/recombinant), data regarding immunosuppression (Human Immunodeficiency Virus, active cancer, high-dose steroids), PHN family history, level of procedure performed, complications, Numeric Rating Scale-11 (NRS-11), Neuropathic Pain Questionnaire (DN4), Short Form-12 (SF-12) quality of life index subscores and average daily tramadol (mg/day) consumption before and 1 and 3 months after the procedure were recorded.

Medication Management Patients' gabapentinoids and antidepressants (amiltriptyline, duloxetine, etc.) used for PHN were continued. Tramadol doses were either increased or decreased for pain control after SPSIPB. Total daily average tramadol consumption was recorded before, at the end of the first and third months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years of age

- who underwent a single-session ultrasound (US)-guided serratus posterior superior intercostal plane block (SPSIPB) in the thoracic region (T1-T10 dermatomes) for PHN between June 2023 and February 2025 were evaluated. -SPSIPB was performed in patients whose complaints persisted despite existing medical treatments.

Exclusion Criteria:Patients were excluded if they had cervical disc herniation -a history of trauma or surgery involving the neck, shoulder, or back; -malignancy- kyphoscoliosis; a history of inflammatory diseases (e.g., rheumatoid arthritis, ankylosing spondylitis)

* congenital anomalies of the spine; neck pain accompanied by neurological deficits
* pregnancy
* mental or psychotic disorders
* hematologic diseases causing bleeding or coagulation disorders
* use of antiplatelet or anticoagulant drugs or other medications predisposing to bleeding
* severe systemic infections such as sepsis
* local infection at the planned intervention site
* known allergy to any of the drugs to be used; or a history of invasive procedures for PHN in the thoracic region within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who underwent a single-session ultrasound (US )guided serratus posterior superior intercostal plane block (SPSIPB) in the thoracic region (T1-T10 dermatomes) for PHN between June 2023 and February 2025 were evaluated. SPSIPB was performed in patients whose complaints persisted despite existing medical treatments.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale -11 (NRS-11) | 3 months
  It is an 11-point scale used to describe pain. It is based solely on the patient's ability to perform activities of daily living and can be used for adults and children ages 10 and older.

SECONDARY OUTCOMES:
Douleur Neuropathique en 4 Questions(DN4) | 3 months
  The DN4 questionnaire is a validated clinical screening instrument designed to detect the presence of neuropathic pain. It was developed by the French Neuropathic Pain Group to address diagnostic challenges and the lack of consensus regarding the identification of neuropathic pain. Owing to its clarity and ease of use, the instrument has been widely adopted in clinical practice and research since 2005.
  The questionnaire comprises four sections and ten individual items. Seven items pertaining to pain quality-including sensory descriptors-are obtained through a structured patient interview and reflect the subjective characteristics of the pain experience. The remaining three items are derived from the clinical examination, during which the clinician evaluates for decreased sensitivity to light touch or pinprick (hypoesthesia), as well as the presence of pain provoked or exacerbated by gentle brushing (allodynia).
Short Form- 12 | 3 months
  The SF-12 consists of 12 items grouped into eight subscales: physical functioning (2 items), role physical (2 items), bodily pain (1 item), general health (1 item), vitality (1 item), social functioning (1 item), role emotional (2 items), and mental health (2 items). Items pertaining to physical and emotional role limitations are dichotomous (yes/no), whereas the remaining items are rated on Likert-type scales ranging from three to six response options.
  The Physical Component Summary (PCS-12) score is derived from the general health, physical functioning, role physical, and bodily pain subscales. The Mental Component Summary (MCS-12) score is calculated from the social functioning, role emotional, mental health, and vitality subscales. Both PCS-12 and MCS-12 scores range from 0 to 100, with higher scores indicating better health status. The SF-12 is a validated and psychometrically robust instrument.

CONTACTS AND LOCATIONS:
Overall Officials: halil ibrahim altun, Principal Investigator — Kanuni Sultan Süleyman Training and Research Hospital
Locations (1):
- İKanuni Sultan Süleyman Training and Research Hospital, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided